CLINICAL TRIAL: NCT03225027
Title: Study on Communication Comprehension in the Schizophrenic Spectrum
Acronym: SKYPROVERB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHRD0814
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia Simple
Keywords: Emotional prosody, schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Gene Expression; Psychiatric Status Rating Scales

STUDY DESIGN:
Intervention Model Description: One experimental procedure proposed to three groups of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with schizophrenia (Experimental): Emotional judgment task, post-experimental questionnaire, recognition task, detection task, questionnaire CAPE-42, trait emotional intelligence questionnaire and positive and negative syndrome scale.
  Interventions: Behavioral: Emotional judgment task; Behavioral: Post-experimental questionnaire; Behavioral: Recognition task; Behavioral: Detection task; Other: CAPE-42; Diagnostic Test: Trait Emotional Intelligence Questionnaire; Diagnostic Test: Positive And Negative Syndrome Scale
- Few psychotic experiences (Experimental): Healthy participants with few psychotic experience. Participants with the lowest score to the CAPE-42 test. Mini International Neuropsychiatric Interview
  Interventions: Behavioral: Emotional judgment task; Behavioral: Post-experimental questionnaire; Behavioral: Recognition task; Behavioral: Detection task; Other: CAPE-42; Diagnostic Test: Trait Emotional Intelligence Questionnaire; Other: Mini International Neuropsychiatric Interview
- Several psychotic experiences (Experimental): Healthy participants with several psychotic experiences. Participants with the highest score to the CAPE-42 test. Mini International Neuropsychiatric Interview
  Interventions: Behavioral: Emotional judgment task; Behavioral: Post-experimental questionnaire; Behavioral: Recognition task; Behavioral: Detection task; Other: CAPE-42; Diagnostic Test: Trait Emotional Intelligence Questionnaire; Other: Mini International Neuropsychiatric Interview

INTERVENTIONS:
Behavioral: Emotional judgment task — Participants had to indicate on a computer the emotional intensity of audio recordings.
Behavioral: Post-experimental questionnaire — Participants will be invited to give us the cognitive strategy used to resolve the emotional judgment task.
Behavioral: Recognition task — Participants will be invited to indicate which recordings they had heard during the emotional judgment task to verify that they have paid attention to the emotional task.
Behavioral: Detection task — Participants indicate every time they heard a given sound in order to verify their audition level.
Other: CAPE-42 — This questionnaire allows evaluating the nature of psychotic experiences.
Diagnostic Test: Trait Emotional Intelligence Questionnaire — To evaluate their emotional intelligence.
  Other Names: TEIQUE
Diagnostic Test: Positive And Negative Syndrome Scale — Evaluating the clinical status of patients with schizophrenia.
  Other Names: PANSS
  Arms: Patients with schizophrenia
Other: Mini International Neuropsychiatric Interview — Evaluating the exclusion criteria in healthy participants.
  Other Names: MINI
  Arms: Few psychotic experiences; Several psychotic experiences

SUMMARY:
The purpose of the present study is to evaluate the effect of emotional prosody on the perception of emotional discourse in the schizophrenic spectrum. The investigators hypothesize that participant may use emotional prosody as an emotional cue to understand the emotional content of discourse.

DETAILED DESCRIPTION:
The integration of ortholinguistic and paralinguistic functions in language, particularly of the emotional prosody, is necessary to interact adaptively with others. People in the schizophrenic spectrum have social difficulties. Is emotional prosody comprehension altered in these people? According to Edwards et al. (2002), there is methodological issues concerning the tasks used to answer this question. Investigators built an emotional judgment task more adapted to study the perception of emotional prosody in the schizophrenic spectrum than the classical paradigm designed to evaluate participants with cerebral injury. The investigators have elaborated a material that consists of 140 short sentences (7±2 words) with a simple syntactic structure. The verbal content expressed positive, neutral or negative emotions. These sentences were announced by four professional actors (two female) with an emotional prosody content congruent or inconsistent with the verbal content. Participants will have to evaluate the emotional intensity of the recordings on a five points Likert scale, from strongly negative to strongly positive. Psychotic experiences of all participants will be evaluated too.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of schizophrenia and being in a stable phase of the disease
* Having between 18 to 60 years old
* Speak french or using french at school
* Accepting not to use psychoactive substances during the preceding 48h
* Being affiliated to the French social security
* Providing their written informed consent

Non-inclusion Criteria:

* Having not audio deficits, nor visual uncorrected deficits
* Having not suffering from depressive symptoms during the last 6 months

Exclusion Criteria:

- Having no neurological, nor psychiatric disease except schizophrenia for the patients groups.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Behavioural measures (response rate and time) | During the experiment
  Participants will have to judge the emotional intensity of audio recordings. In this task, the participant is asked to judge the emotional intensity of audio recordings of men and women (2 actors + 2 actresses): he / she must press a button as quickly as possible to indicate whether the Audio recordings presented via small speakers are very negative, negative, non-emotional, positive or very positive (5 possible choices).
  The response time variable may be added as a co-variable in order to avoid perceptive-motor disorders (medication-related and / or general motor slowdown) that may influence the results of time-of- answers.

SECONDARY OUTCOMES:
Symptomatic impact | During the experiment
  Evaluate the nature of the psychotic experiments (CAPE-42 test).
Evaluate the cognitive functioning | During the experiment
  Neuropsychological tests will allow evaluating the cognitive profile of the participants that can impact their behaviour during the experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Mouna TRABELSI, MD, Principal Investigator — HDJ François Villon (Centre Hospitaliser René-Dubos); Virginie BEAUCOUSIN, PhD, Study Chair — CRFDP (University of Rouen)
Locations (1):
- HDJ François Villon, Cergy-Pontoise, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brazo P, Beaucousin V, Lecardeur L, Razafimandimby A, Dollfus S. Social cognition in schizophrenic patients: the effect of semantic content and emotional prosody in the comprehension of emotional discourse. Front Psychiatry. 2014 Sep 10;5:120. doi: 10.3389/fpsyt.2014.00120. eCollection 2014. PMID 25309458
- [Result] Edwards J, Jackson HJ, Pattison PE. Emotion recognition via facial expression and affective prosody in schizophrenia: a methodological review. Clin Psychol Rev. 2002 Jul;22(6):789-832. doi: 10.1016/s0272-7358(02)00130-7. PMID 12214327
- [Result] Beaucousin V, Lacheret A, Turbelin MR, Morel M, Mazoyer B, Tzourio-Mazoyer N. FMRI study of emotional speech comprehension. Cereb Cortex. 2007 Feb;17(2):339-52. doi: 10.1093/cercor/bhj151. Epub 2006 Mar 8. PMID 16525130